CLINICAL TRIAL: NCT02184013
Title: Correlation of Arrhythmia Mechanism and Substrate to Ablate Persistent Atrial Fibrillation:A Pilot Study
Brief Title: Correlation of the Arrhythmia Mechanism and Substrate to Ablate Persistent Atrial Fibrillation Study
Acronym: COAST-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140623
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Delayed gadolinium enhanced MRI; C-metahydroxyepherdrine (HED) PET scan; ECGI mapping; Atrial Fibrosis; Atrial sympathetic denervation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation (in addition ot PVI) guided by ECGI mapping, and atrial fibrosis mapping (DE-MRI).

SUMMARY:
This is a pilot study to assess the usefulness of ECG mapping, and enhanced MRI and PET scan imaging in identifying atrial fibrosis and arrhythmia circuits involved in persistent atrial fibrillation and in guiding an innovative AF catheter ablation strategy.

It is hypothesized that identifying these critical arrhythmia circuits and atrial fibrosis with enhanced imaging and performing an individualized innovative AF catheter ablation will result in higher procedural success rates.

DETAILED DESCRIPTION:
Pulmonary vein isolation catheter ablation for the treatment of persistent AF (PeAF)or longstanding persistent AF is associated with success rates of 40-50% at one year. Experimental models have shown that AF results in progressive structural changes due to electrical atrial remodeling, where AF burden correlates with atrial fibrosis. The optimal ablation strategy for patients with PeAF is not yet known. There is limited understanding of the critical mechanisms responsible for maintenance of AF in these patients.

In this study ECG body mapping (ECGI) will be used to look for distinct electrical rotors in the atria. Delayed gadolinium enhanced magnetic resonance imaging (DE-MRI) will be used to assess the extent of left atrial fibrosis. In addition to PVI catheter ablation procedure, an ablation strategy guided by the results of the ECGI mapping and DE-MRI will be performed.A C-metahydroxyepherdrine (HED) PET scan will also be done pre-ablation to evaluate left atrial sympathetic denervation and any relationship to the initiation and/or maintenance of AF.

Subjects will be seen at 3 and 6 months after ablation, with 12 lead ECG and 2-week loop monitoring done at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤ 80 years;
* Symptomatic persistent AF AND clinically indicated for AF catheter ablation
* At least one episode of AF lasting more than 7 days, documented on 12-lead ECG, Holter monitor, 2-week loop monitor or trans-telephonic monitor (TTM) within 12 months of enrollment in the study
* Able to provide informed consent.

Exclusion Criteria:

* History of previous catheter or surgical ablation for AF
* Presence of intracardiac thrombus
* contraindication to systemic oral anticoagulation therapy
* Subjects with reversible causes of AF
* Antero-posterior left atrial dimension > 60 mm on echocardiography
* Severe valvular disease (mitral/aortic stenosis or regurgitation);
* Subjects that are pregnant or breastfeeding;
* Chronic kidney disease and creatinine clearance <50ml/min.
* Contraindication to MRI Imaging (e.g. permanent pacemaker, metallic implants, etc)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation (AF) Termination | During catheter ablation
  AF termination resulting in restoration of sinus rhythm during ablation.

SECONDARY OUTCOMES:
Radio frequency (RF) ablation time | During catheter ablation
Procedure Duration | During catheter ablation
  Total procedure duration
Freedom from AF | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pablo B Nery, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Robert deKemp, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation; Elena Pena, MD, Principal Investigator — The Ottawa Hospital; David H Birnie, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada